CLINICAL TRIAL: NCT06386705
Title: A Multicenter, Open-label, Phase Ia/Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of TSN084 Tablets in Patients With Advanced Malignant Tumors.
Brief Title: TSN084 Treating Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tyligand Bioscience (Shanghai) Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSN084-101CH
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Phase 1a (Experimental): Dose Escalation/Evaluation
  Interventions: Drug: TSN084
- Experimental: Phase 1b (Experimental): TSN084 recommended Phase 2 dose administered to separate cohorts of patients with selected malignancies harboring mutations including but not limited to MET exon14 skipping mutation and MET amplification.
  Interventions: Drug: TSN084

INTERVENTIONS:
Drug: TSN084 — TSN084 will be administered at the assigned dose level, orally, until disease progression or intolerable toxicity.

SUMMARY:
TSN084 is a novel type II kinase inhibitor with demonstrated anti-tumor effects in vitro and in vivo and targets multiple tyrosine kinases, such as c-MET, FLT3, TRK and serine/threonine kinase CDK8/19. This phase 1a/1b study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of TSN084 in advanced or metastatic malignancies in China.

DETAILED DESCRIPTION:
The phase 1a part will begin with an exploration of TSN084 dose and regimen to determine the maximum tolerated dose (MTD) and/or recommended dose for further investigation (i.e., RP2D). In Phase 1b part, separate cohorts of patients with different histological diagnosis will be evaluated for the clinical activity and efficacy of TSN084 at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old.
* The subject fully understands the requirements of the study and voluntarily signs the written informed consent.
* Be able to comply with the medication requirements of the study and all study related procedures and evaluations; not deemed as potentially unreliable and/or uncooperative.
* Meeting the requirements of tumor types shown below. Phase Ia Study: Histological or cytological diagnosis of locally advanced, relapsed, or metastatic malignancies, not amenable to standard therapy or for which no standard therapy is available.

Phase Ib study: Histological or cytological diagnosis of the locally advanced, relapsed, or metastatic selected malignancies not amenable to standard therapy (disease progression or intolerance), or unable to receive standard therapy/no standard therapy is available. Malignancies with targeted mutations are preferred, including but not limited to MET exon 14 skipping mutation and MET amplification.

* Survival expectations are ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 for Phase Ia, while 0 to 2 for Phase Ib.
* Patients with adequate organ function at the time of screening.
* Male and female patients of childbearing potential must agree to use effective methods of contraception.

Exclusion Criteria:

* Patients with active brain metastases, except that their central nervous system (CNS) tumor metastases are confined to the supratentorial or cerebellum, have been adequately treated (surgery or radiotherapy), have maintained radiographic stability for at least 4 weeks, and do not require corticosteroids to control symptoms.
* Other malignancies (other than non-melanoma basal cell carcinoma or squamous cell carcinoma of the skin, breast/cervical carcinoma in situ, superficial bladder carcinoma that have received radical treatment and no evidence of disease recurrence) within 5 years prior to initiation of TSN084 treatment;
* Any arterial thromboembolic event, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred within 6 months prior to enrolment;
* Uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (Patients who do not need drainage effusion or have no significant increase in effusion after 3 days of cessation of drainage can be included).
* Has active gastrointestinal disease or other disease, or other factors such as surgical resection that may significantly affect drug absorption, metabolism, or excretion.
* Pregnant or lactating women.
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* HIV infected patients (HIV 1/2 antibody positive).
* Known active syphilis infection, or active tuberculosis.
* A history of drug abuse or drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days
  Number of patients with dose limiting toxicity, to determine the MTD and/or RP2D
Incidence of Treatment-Emergent Adverse Events (TEAE) | Up to 3 years
  Incidence of TEAE, Serious Adverse Event (SAE), their relationship with the investigational product and severity. Adverse events will be graded according to NCI-CTCAE V5.0.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
  To characterize the pharmacokinetic (PK) properties of TSN084 in patients with advanced malignant tumors.
Time to Cmax (Tmax) | 28 days
  To characterize the pharmacokinetic (PK) properties of TSN084 in patients with advanced malignant tumors.
Area under the concentration versus time curve from time 0 to the last measurable concentration (AUC 0-t) | 28 days
  To characterize the pharmacokinetic (PK) properties of TSN084 in patients with advanced malignant tumors.
Objective response rate (ORR) | Up to 3 years
  Tumor response assessments by RECIST v1.1
Duration of response (DoR) | Up to 3 years
  Tumor response assessments by RECIST v1.1
Disease control rate (DCR) | Up to 3 years
  Tumor response assessments by RECIST v1.1
Time to response (TTR) | Up to 3 years
  Tumor response assessments by RECIST v1.1
Progression free survival (PFS) | Up to 3 years
  Tumor response assessments by RECIST v1.1
Overall survival (OS) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking university cancer hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No